CLINICAL TRIAL: NCT07088575
Title: Practice of Deep Venous Thrombosis Prophylaxis and Its Incidence in Patients Undergoing Gastrointestinal and Hepatobiliary Surgery: A Nepalese Single-center, Retrospective Study
Brief Title: Practice of Deep Venous Thrombosis Prophylaxis and Its Incidence in Patients Undergoing Gastrointestinal and Hepatobiliary Surgery
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Prajjwol Luitel, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 589(6-11)E2.079/080
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients >18 years who underwent major gastrointestinal or hepatobiliary surgery
  Interventions: Procedure: major gastrointestinal or hepatobiliary surgery under general anesthesia

INTERVENTIONS:
Procedure: major gastrointestinal or hepatobiliary surgery under general anesthesia — major gastrointestinal or hepatobiliary surgery under general anesthesia

SUMMARY:
Recent studies from Asia have reported a wide variation in the incidence of deep vein thrombosis (DVT), ranging from 5% to 50% in patients undergoing major abdominal surgery. However, data specific to the Nepalese population remains unavailable. This study aims to evaluate current thromboprophylaxis practices and determine the incidence of DVT in Nepalese adults undergoing gastrointestinal and hepatobiliary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years
* Underwent major gastrointestinal or hepatobiliary surgery
* Surgery performed under general anesthesia
* Major surgery defined as any operative intervention in the abdominal or hepatobiliary region requiring general anesthesia

Exclusion Criteria:

* History of VTE within 3 months before surgery
* Known hypercoagulable state or congenital thrombophilia
* Diagnosis of atrial fibrillation
* Undergoing systemic cancer chemotherapy or radiotherapy within the past 15 days
* Pregnant or lactating women
* Missing information in clinical records
* Non-operated patients or those receiving conservative management
* Patients undergoing liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients aged >18 years who underwent major gastrointestinal or hepatobiliary surgery under general anesthesia at a tertiary referral center in Nepal. Patients were identified retrospectively through departmental audit records from the Department of Surgical Gastroenterology between October 2021 and April 2024. Major surgery was defined as any operative intervention involving the abdominal or hepatobiliary region requiring general anesthesia. Surgical procedures were categorized by organ system into upper gastrointestinal, hepatopancreatobiliary (HPB), colorectal, and other (e.g., small intestine, retroperitoneum, abdominal wall). Patients with a recent history of venous thromboembolism (VTE), known hypercoagulable conditions, atrial fibrillation, ongoing cancer therapy, pregnancy, or incomplete clinical data were excluded from the study. Data collected included demographic, clinical, intraoperative, and postoperative variables relevant to thromb
Sampling Method: Non-Probability Sample
Enrollment: 1530 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Use of Thromboprophylaxis and Incidence of DVT in Major GI and Hepatobiliary Surgeries | From date of surgery until hospital discharge or up to 30 days postoperatively, whichever occurs first
  This outcome assesses the proportion of patients receiving appropriate thromboprophylaxis, as well as the incidence of deep vein thrombosis (DVT) among individuals undergoing major gastrointestinal and hepatobiliary surgeries. Data will be collected to evaluate adherence to prophylaxis guidelines and to determine the effectiveness of thromboprophylactic measures in preventing DVT in this surgical population.

CONTACTS AND LOCATIONS:
Overall Officials: Prajjwol Luitel, MBBS, Principal Investigator — Maharajgunj Medical Campus
Locations (1):
- Maharajgunj Medical Campus, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to demographic characteristics, surgical details, thromboprophylaxis use, and DVT outcomes will be shared. This includes preoperative, intraoperative, and postoperative variables as collected in the study.
Supporting Information: SAP, Analytic Code
Time Frame: The IPD and supporting documents will be available beginning six months after publication of the study results and will remain available for up to five years thereafter.
Access Criteria: Access will be granted to qualified researchers and institutions conducting ethically approved research. Requests must include a brief study proposal and intended use. Data will be made available through a secure data-sharing platform upon signing a data use agreement.